CLINICAL TRIAL: NCT03113318
Title: Total Mediastinal Lymph Node Dissection in Pulmonary Metastasectomy From Colorectal Cancer - a Randomized, Controlled Trial
Brief Title: Mediastinal Lymph Node Dissection in Conjunction With Pulmonary Metastasectomy From Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Kåre Hornbech, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Khornbech
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Lung Neoplasms; Neoplasm Metastasis; Colorectal Cancer
Keywords: Pulmonary neoplasm; Metastasis; colorectal neoplasm
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lymph node dissection and pulmonary metastasectomy (Experimental): Total mediastinal lymph node dissection and pulmonary metastasectomy from colorectal cancer
  Interventions: Procedure: Total mediastinal lymph node dissection and pulmonary metastasectomy
- Pulmonary metastasectomy only (Active Comparator): Only pulmonary metastasectomy from colorectal cancer
  Interventions: Procedure: Only pulmonary metastasectomy

INTERVENTIONS:
Procedure: Total mediastinal lymph node dissection and pulmonary metastasectomy — Total mediastinal lymph node dissection where all lymph nodes and fatty tissues is removed conjunction with pulmonary metastasectomy
  Arms: Lymph node dissection and pulmonary metastasectomy
Procedure: Only pulmonary metastasectomy
  Arms: Pulmonary metastasectomy only

SUMMARY:
To study whether or not total mediastinal lymph node dissection in conjunction with pulmonary metastasectomy from colorectal cancer is associated with improved survival compared to pulmonary metastasectomy only.

DETAILED DESCRIPTION:
The question of lymph node sampling and/or involvement in pulmonary metastasectomy remains controversial. The performance of lymph node dissection during pulmonary metastasectomy is infrequent and varies between institutions. Of all the patients in The International Registry of Lung Metastases only 4,6% of patients underwent lymph node dissection. In a recent survey by Internullo and colleagues amongst the members of European Society of Thoracic Surgeons 55% perform mediastinal lymph node sampling whereas 33% perform no nodal sampling at all. The rate of lymph node involvement varies between primary tumours.

Several studies from groups that systematically perform mediastinal lymph node dissection in conjunction with pulmonary metastasectomy have been published and in all studies the presence of lymph node metastasis emerges as an ominous prognostic factor. Ercan and colleagues found a 3-year survival of 69% for patients without lymph node involvement versus 38% in patients with positive lymph nodes. Saito and colleagues reported a 5-year survival of 53,6 for patients without hilar or mediastinal node involvement versus 6,2% at 4 years for patients with positive nodes. Bölükbas and colleagues reported a 5-year survival of 59% for patients without lymph node involvement in contrast to 23% for patients with lymph node involvement.

The rate of lymph node involvement is reported between 20-43% and risk factors for lymph node involvement include 2 or more metastases, prior liver metastases, rectum cancer and size of metastases .

Most of the above mentioned authors are in favor of mediastinal lymphadenectomy but also stress that the evidence available is not solid enough to make firm recommendations. In conclusion the literature is quite limited and of low-level evidence.

In remains unclear whether the complete removal of mediastinal lymph nodes is associated with a survival benefit or merely allows for a more accurate postoperative staging and guidance for additional oncological treatment. Thus, the aim of the following proposed study is to examine whether or not systemic lymph node dissection during pulmonary metastasectomy is associated with a survival benefit.

Hypothesis:

1. Systemic mediastinal lymphadenectomy during pulmonary metastasectomy with curative intent for colorectal carcinoma (CRC) is feasible and safe.
2. Systemic mediastinal lymphadenectomy during pulmonary metastasectomy with curative intent for CRC is associated with improved survival compared to only pulmonary metastasectomy.

Design:

Prospective, randomized, controlled trial. No lymph node dissection versus systemic mediastinal lymph node dissection with en-bloc resection of lymph nodes and fatty tissue in station 2,4,7,8, 9 and 10 on the right side and 5,6,7,8, 9 and 10 on the left side during pulmonary metastasectomy for CRC.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Able to give informed consent
* Willing to be randomized

Exclusion Criteria:

* Previous mediastinal lymphadenectomy
* Previous pulmonary metastasectomy
* Evidence of other metastasetic disease
* Primary tumor is not under control
* Five metastases or more
* If final histologic examination of the resected lung lesion(s) reveals other histology than colorectal metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 7-8 years

SECONDARY OUTCOMES:
1-year overall survival | 3-4 years
3-year overall survival | 4-5 years
1-, 3-, 5-year disease free survival | 7-8 years
Number of lymph nodes removed | 2-3 years
30- day morbidity | 2-3 years
30-day mortality | 2-3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Internullo E, Cassivi SD, Van Raemdonck D, Friedel G, Treasure T; ESTS Pulmonary Metastasectomy Working Group. Pulmonary metastasectomy: a survey of current practice amongst members of the European Society of Thoracic Surgeons. J Thorac Oncol. 2008 Nov;3(11):1257-66. doi: 10.1097/JTO.0b013e31818bd9da. PMID 18978560
- [Background] Ercan S, Nichols FC 3rd, Trastek VF, Deschamps C, Allen MS, Miller DL, Schleck CD, Pairolero PC. Prognostic significance of lymph node metastasis found during pulmonary metastasectomy for extrapulmonary carcinoma. Ann Thorac Surg. 2004 May;77(5):1786-91. doi: 10.1016/S0003-4975(03)01200-1. PMID 15111187
- [Background] Saito Y, Omiya H, Kohno K, Kobayashi T, Itoi K, Teramachi M, Sasaki M, Suzuki H, Takao H, Nakade M. Pulmonary metastasectomy for 165 patients with colorectal carcinoma: A prognostic assessment. J Thorac Cardiovasc Surg. 2002 Nov;124(5):1007-13. doi: 10.1067/mtc.2002.125165. PMID 12407386
- [Background] Bolukbas S, Sponholz S, Kudelin N, Eberlein M, Schirren J. Risk factors for lymph node metastases and prognosticators of survival in patients undergoing pulmonary metastasectomy for colorectal cancer. Ann Thorac Surg. 2014 Jun;97(6):1926-32. doi: 10.1016/j.athoracsur.2014.02.026. Epub 2014 Mar 28. PMID 24681037
- [Background] Renaud S, Alifano M, Falcoz PE, Magdeleinat P, Santelmo N, Pages O, Massard G, Regnard JF. Does nodal status influence survival? Results of a 19-year systematic lymphadenectomy experience during lung metastasectomy of colorectal cancer. Interact Cardiovasc Thorac Surg. 2014 Apr;18(4):482-7. doi: 10.1093/icvts/ivt554. Epub 2014 Jan 16. PMID 24442624